CLINICAL TRIAL: NCT00786188
Title: A Phase 2, Exploratory, Eight-Week, Multicenter, Double-Blind, Randomized, Placebo-Controlled, Efficacy and Safety Study of Mesafem (Paroxetine Mesylate) Capsules in the Treatment of Vasomotor Symptoms Associated With Menopause
Brief Title: Eight-Week Efficacy & Safety Study of Brisdelle™ (Formerly Known as Mesafem) in the Treatment of Vasomotor Symptoms Associated With Menopause
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Noven Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N30-002
Record Dates: First submitted 2008-11-04; First posted 2008-11-06 (Estimated); Results first posted 2014-03-12 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Hot Flashes
Keywords: Menopause; Vasomotor Symptoms; Hot flash; Perimenopause; Nonhormonal therapies; Climacteric symptoms; Mesafem; Low-Dose Mesylate salt of Paroxetine (LDMP)
MeSH Terms: conditions — Hot Flashes | interventions — Paroxetine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brisdelle (paroxetine mesylate) (Experimental): Eligible subjects will be randomized to receive Brisdelle (paroxetine mesylate) Capsules 7.5 mg.
  Interventions: Drug: Brisdelle (paroxetine mesylate)
- Placebo - Sugar Pill (Placebo Comparator): Eligible subjects will be randomized to receive a sugar pill.
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Brisdelle (paroxetine mesylate) — Eligible subjects will be randomized to receive Brisdelle™ (paroxetine mesylate) Capsules 7.5 mg.
  Other Names: Former Names: Mesafem capsules 7.5 mg or; LDMP (Low-Dose Mesylate salt of Paroxetine)
  Arms: Brisdelle (paroxetine mesylate)
Drug: Sugar pill — Subjects will receive a sugar pill.
  Arms: Placebo - Sugar Pill

SUMMARY:
This is an exploratory 8-week, multicenter, double-blind, randomized, placebo-controlled study of Brisdelle (paroxetine mesylate) Capsules 7.5 mgin subjects with moderate to severe postmenopausal vasomotor symptoms (VMS), defined as follows:

* Moderate VMS: Sensation of heat with sweating, able to continue activity
* Severe VMS: Sensation of heat with sweating, causing cessation of activity

DETAILED DESCRIPTION:
Eligible subjects will be entered into a 1-week observation period followed by a 1-week run-in period. Following completion of the run-in period, eligible subjects will be randomized to receive either Brisdelle (paroxetine mesylate) Capsules 7.5 mg or placebo in a 1:1 ratio. Study drug will be administered once daily at bedtime. Symptom assessment questionnaires will be administered at baseline and at Day 28 and Day 57 visits.

ELIGIBILITY:
Inclusion Criteria:

1. Female, >40 years of age
2. Reported more than 7-8 moderate to severe hot flashes per day (average) or 50-60 moderate to severe hot flashes per week for at least 30 days prior
3. Spontaneous amenorrhea for at least 12 consecutive months
4. Amenorrhea for at least 6 months and meet the biochemical criteria for menopause
5. Bilateral salpingo-oophorectomy >6 weeks with or without hysterectomy

Exclusion Criteria:

1. History of hypersensitivity or adverse reaction to paroxetine mesylate
2. Use of an investigational study medication within 30 days prior to screening or during the study
3. Concurrent participation in another clinical trial or previous participation in this trial
4. Family of investigational-site staff

Min Age: 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick F. Freuen, MD, Principal Investigator — North Spokane Women's Clinic, Spokane, WA 99207; Richard E. Hedrick, MD, Principal Investigator — Hawthorne Medical Research, Inc., Winston-Salem, NC 27103; Samuel N. Lederman, MD, Principal Investigator — Altus Research, Lake Worth, FL 33461; Larry S. Seidman, DO, Principal Investigator — Philadelphia Clinical Research, LLC, Philadelphia, PA 19114; James E. Tomblin, MD, Principal Investigator — Hawthorne Medical Research, Inc., Greensboro, NC 27408; Peter A. Zedler, MD, Principal Investigator — Virginia Women's Center, Richmond, VA 23233; D. S. Harnsberger, MD, Principal Investigator — Chattanooga Medical Research, LLC, Chattanooga, TN 37404; John A. Hoekstra, MD, Principal Investigator — National Clinical Research, Inc., Richmond, VA 23294; Robin Kroll, MD, Principal Investigator — Women's Clinical Research Center, Seattle, WA 98105; Ashley Tunkle, MD, Principal Investigator — Anchor Research Center, Naples, FL 34102
Locations (10):
- United States (10):
  - Altus Research, Lake Worth, Florida
  - Anchor Research Center, Naples, Florida
  - Hawthorne Research, Greensboro, North Carolina
  - Hawthorne Medical Research, Inc., Winston-Salem, North Carolina
  - Philadelphia Clinical Research, Philadelphia, Pennsylvania
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - Virginia Women's Center, Richmond, Virginia
  - National Clinical Research, Inc., Richmond, Virginia
  - Women's Clinical Research Center, Seattle, Washington
  - North Spokane Women's Clinic Research, Spokane, Washington

REFERENCES:
- [Background] Fugate SE, Church CO. Nonestrogen treatment modalities for vasomotor symptoms associated with menopause. Ann Pharmacother. 2004 Sep;38(9):1482-99. doi: 10.1345/aph.1D610. Epub 2004 Aug 3. PMID 15292498
- [Background] Kritz-Silverstein D, Goldani Von Muhlen D, Barrett-Connor E. Prevalence and clustering of menopausal symptoms in older women by hysterectomy and oophorectomy status. J Womens Health Gend Based Med. 2000 Sep;9(7):747-55. doi: 10.1089/15246090050147727. PMID 11025867
- [Background] Nelson HD, Vesco KK, Haney E, Fu R, Nedrow A, Miller J, Nicolaidis C, Walker M, Humphrey L. Nonhormonal therapies for menopausal hot flashes: systematic review and meta-analysis. JAMA. 2006 May 3;295(17):2057-71. doi: 10.1001/jama.295.17.2057. PMID 16670414
- [Background] Greene JG. A factor analytic study of climacteric symptoms. J Psychosom Res. 1976;20(5):425-30. doi: 10.1016/0022-3999(76)90005-2. No abstract available. PMID 1003364

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period = 29 October 2008 to 26 May 2009 Types of Locations = Research clinics
Pre-assignment Details: Eligible subjects were entered into a 1-week observation period followed by a 1-week run-in period. After completion of run-in period, eligible subjects were randomized to receive either Brisdelle (paroxetine mesylate) Capsules 7.5 mg or placebo in a 1:1 ratio. Study drug was administered once daily at bedtime.
Groups:
- Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg: Interventions Administered:
  Subjects received Brisdelle (paroxetine mesylate) Capsules 7.5 mg administered once daily at bedtime.
  Eligible subjects were entered into a 1-week observation period followed by a 1-week run-in period. After completion of run-in period, eligible subjects were randomized to receive Brisdelle (paroxetine mesylate) Capsules 7.5 mg administered once daily at bedtime.
- Placebo - Sugar Pill: Interventions Administered:
  Subjects received placebo capsules administered once daily at bedtime.
  Eligible subjects were entered into a 1-week observation period followed by a 1-week run-in period. After completion of run-in period, eligible subjects were randomized to receive placebo administered once daily at bedtime.
Period: Overall Study
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg | Placebo - Sugar Pill
Started | 50 | 52
Completed | 45 | 51
Not Completed | 5 | 1
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg: Eligible subjects will be randomized to receive Brisdelle (paroxetine mesylate) Capsules 7.5 mg.
- Total: Total of all reporting groups
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg | Placebo - Sugar Pill | Total
Number analyzed (Participants) | 50 | 52 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 49 | 95
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (55.8) | 55.0 (54.6) | 55.0 (55.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 52 | 102
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 52 | 102

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Hot Flash Frequency at Week 4 and Week 8
Description: The number of hot flashes reported in the result table are:
  * Mean change in frequency of moderate to severe VMS from baseline to Week 4
  * Mean change in frequency of moderate to severe VMS from baseline to Week 8. They are both measured as hot flashes per week.
Time Frame: Week 4 and Week 8
Population: MODIFIED ITT (MITT) POPULATION Brisdelle 49 (98.0%) Placebo 52 (100.0%) PER PROTOCOL (PP) POPULATION Brisdelle 45 (90.0%) Placebo 51(98.1%)
Measure: Mean (Standard Error); unit: Hot flashes
Groups:
- Brisdelle (Paroxetine Mesylate) Capsules: Eligible subjects will be randomized to receive Brisdelle (paroxetine mesylate) Capsules 7.5 mg capsules.
  Subjects will be randomized to one of the two treatments in a 1:1 ratio
- Placebo - Sugar Pill: Eligible subjects will be randomized to receive a sugar pill. Subjects will be randomized to one of the two treatments in a 1:1 ratio.
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo - Sugar Pill
Number analyzed (Participants) | 49 | 52
Hot flashes
  Baseline | 82.44 (3.14) [0 to 0] | 83.18 (3.67) [0 to 0]
  Week 4 | 37.3 (3.11) [-15.70 to -1.92] | 28.5 (3.30) [-15.70 to -1.92]
  Week 8 | 42.2 (3.24) [-13.52 to 0.16] | 35.5 (3.13) [-13.52 to 0.16]
Statistical Analysis 1: Comparison: Brisdelle (Paroxetine Mesylate) Capsules vs Placebo - Sugar Pill; Test type: Superiority or Other; p = 0.0177, Repeated measures analysis — Week 4 frequency
Statistical Analysis 2: Comparison: Brisdelle (Paroxetine Mesylate) Capsules vs Placebo - Sugar Pill; Test type: Superiority or Other; p = 0.0541, Reapeated measures analysis — Week 8 frequency

2. Primary Outcome: Mean Change From Baseline in Hot Flash Severity at Week 4 and Week 8
Description: A scale was not used to measure severity scores. Severity scores of hot flashes were calculated for each subject. The following formula was used to calculate severity.
  SS = (2•Fm + 3•Fs) ÷ (Fm + Fs)
  Where:
  SS = severity score Fm = frequency of moderate hot flashes Fs = frequency of severe hot flashes The mean number of moderate and severe hot flashes that was recorded in the Run-In Period was used to calculate the baseline severity score.
Time Frame: Week 4 and Week 8
Measure: Mean (Standard Error); unit: Severity score
Groups:
- Brisdelle (Paroxetine Mesylate) Capsules: Eligible subjects will be randomized to receive Brisdelle (paroxetine mesylate) Capsules 7.5 mg. Subjects will be randomized to one of the two treatments in a 1:1 ratio.
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo - Sugar Pill
Number analyzed (Participants) | 48 | 51
Severity score
  Baseline | 2.570 (0.044) | 2.539 (0.035)
  Week 4 | 0.128 (0.031) | 0.072 (0.024)
  Week 8 | 0.133 (0.032) | 0.066 (0.026)
Statistical Analysis 1: Comparison: Brisdelle (Paroxetine Mesylate) Capsules vs Placebo - Sugar Pill; Test type: Superiority or Other; p = 0.0644, Reapeated measures analysis — Week 4 severity
Statistical Analysis 2: Comparison: Brisdelle (Paroxetine Mesylate) Capsules vs Placebo - Sugar Pill; Test type: Superiority or Other; p = 0.0364, Reapeated measures analysis — Week 8 severity

3. Secondary Outcome: Change From Baseline in Climacteric Symptoms at Week 8
Description: The Greene Climacteric Scale (GCS) was used for this measurement. The scale has 21 questions and measures symptoms in 4 areas; these are psychological (anxiety and depression), physical, vasomotor, and libido.
  The severity of the symptom was scored as: 0=none, 1=mild, 2=moderate, and 3=severe. Anxiety was determined by using the sum of scores 1 to 6, and depression was determined by using the sum of scores 7 to 11. Physical aspects were determined by using the sum of scores 12 to 18; vasomotor aspects were determined by using the sum of scores 19 to 20; and libido was determined by using the score for question 21.
  The total GCS score ranges from "0" to "63" which is the sum of all the scores for the 21-symptom assessment questions in this scale. Each subject's total GCS score at baseline and at Week 8 were used to calculate change from baseline in these symptoms. The change from baseline is reported below.
Time Frame: Week 8
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo - Sugar Pill
Number analyzed (Participants) | 47 | 51
units on a scale
  Baseline | 16.63 (1.55) | 17.33 (1.32)
  Week 8 | 12.31 (9.24) | 12.67 (6.90)

4. Secondary Outcome: Change From Baseline in Hot Flash Composite Score at Week 4 and Week 8
Description: A scale was not used for this measurement.
  Composite scores of hot flashes were calculated by using the following formula:
  CS = (2 • Fm + 3 • Fs)
  Where:
  CS = composite score Fm = frequency of moderate hot flashes Fs = frequency of severe hot flashes The mean number of moderate and severe hot flashes recorded in the Run-In Period was used to calculate the baseline composite score.
Time Frame: Week 4 and Week 8
Measure: Mean (Standard Error); unit: Composite score
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo - Sugar Pill
Number analyzed (Participants) | 48 | 51
Composite score
  Baseline | 211.9 (8.85) | 213.0 (11.34)
  Week 4 | 114.7 (8.43) | 136.4 (9.01)
  Week 8 | 102.6 (8.82) | 119.2 (8.47)

5. Secondary Outcome: Effect of Brisdelle (Paroxetine Mesylate) Capsules on Depression and Anxiety at Week 8
Description: Depression & anxiety were measured using the Hospital Anxiety & Depression Scale (HADS).
  The HADS is a scale developed to assess anxiety & depression. The HADS Scale consists of 14 Questions (7 relating to anxiety; 7 relating to depression) with possible scores ranging from 0 to 21.
  The results presented below are the number of participants with abnormal HADS Scores for both Abnormal Anxiety & Abnormal Depression combined at Week 8.
Time Frame: Week 8
Measure: Number; unit: participants
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo - Sugar Pill
Number analyzed (Participants) | 44 | 50
participants
  Baseline | 2 | 1
  Week 4 | 0 | 1
  Week 8 | 0 | 1

6. Secondary Outcome: Effect of Brisdelle (Paroxetine Mesylate) Capsules on Mood at Week 4
Description: Mood was measured using the Profile of Mood States (POMS) Questionnaire. The Profile of Moods States (POMS) is a 65-item multi-dimensional measure that provides a method of assessing transient, fluctuating active mood states. Key areas that are measured include: tension-anxiety, anger-hostility, fatigue-inertia, depression-dejection, vigor-activity, confusion-bewilderment. Responses to questions are scored with the following numerical values: Not at all = 1, A little = 2, Moderate = 3, Quite a bit = 4, Extremely = 5. A total score for a domain was obtained by summing the responses of individual items in the domain. The total POMS score can range from "65" to "335."
  The percentage of participants who had a change from baseline in the total score at Week 4 is reported below.
Time Frame: Week 4
Measure: Number; unit: percentage of participants
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo - Sugar Pill
Number analyzed (Participants) | 48 | 49
percentage of participants | 21 | 18

7. Secondary Outcome: Effect of Brisdelle (Paroxetine Mesylate) Capsules on Improvement of Hot Flash Interference at Week 4
Description: Interference of hot flashes was measured by using the Hot Flash-Related Daily Interference Scale (HFRDIS). The HFRDIS is a 10-item scale that measures the degree to which hot flashes interfere with 9 daily activities and the tenth item measures the degree to which hot flashes interfere with each of the other items. Subjects can score for each item on a scale from 0 to 10 where 0 = Do not interfere and a score of 10 = Completely interferes.
  The measure being reported below is percentage of responders who had an improvement in HFRDIS score at Week 4 compared to baseline. A responder is defined as a subject who had an improvement in the HFRDIS score. An improvement is define as a score ≤3 on each question.
Time Frame: Week 4
Measure: Number; unit: percentage of responders
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo - Sugar Pill
Number analyzed (Participants) | 46 | 47
percentage of responders | 12 | 11

8. Secondary Outcome: Proportion of Clinical Global Impression (CGI) Responders at Week 4 and Week 8
Description: The Clinical Global Impression Scale (CGIS) was completed by the investigator and was used to measure the severity of the VMS at any given time and the improvement from baseline. Responders were defined as subjects who achieved a score of 1 to 3 where 1 = very much improved, 2 = much improved, and 3 = minimally improved. Non-responders were defined as subjects who achieved a score of 4 to 7 where 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse.
Time Frame: Week 4 and Week 8
Measure: Number; unit: Percentage of participants
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo - Sugar Pill
Number analyzed (Participants) | 46 | 50
Percentage of participants
  Week 4 | 73.91 | 60.00
  Week 8 | 64.58 | 54.90

9. Secondary Outcome: Asses the Effect of Brisdelle (Paroxetine Mesylate) Capsules on the Interference on Sexual Functioning at Week 8
Description: The Arizona Sexual Experiences Scale (ASEX) is a 5-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm. Possible total scores range from 5 to 30, with the higher scores indicating more sexual dysfunction. The sum of the scores for all 5 items was calculated.
Time Frame: Week 8
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo - Sugar Pill
Number analyzed (Participants) | 48 | 49
units on a scale
  Baseline | 17.98 (0.67) | 17.33 (0.72)
  Week 8 | 18.00 (0.90) | 18.15 (1.44)

10. Secondary Outcome: Proportion of Numerical Rating Scale (NRS) True Responders at Week 4 and Week 8
Description: The Subject Impression Numerical Rating Scale (NRS) is an 11-point scale was used to measure how bothered a subject was by hot flashes both during the day and the night.
  The measure being reported below is percentage of responders who had an improvement in NRS score at Week 4 compared to baseline. A responder is defined as a subject who had an improvement in the NRS score. An improvement is define as a score ≤3 on each question.
Time Frame: Week 4 and Week 8
Measure: Number; unit: Percentage of true responders
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo - Sugar Pill
Number analyzed (Participants) | 48 | 49
Percentage of true responders
  Week 4 | 33.33 | 16.67
  Week 8 | 37.14 | 21.95

11. Secondary Outcome: Effect of Brisdelle (Paroxetine Mesylate) Capsules on BMI at Week 4 and Week 8
Description: Body Mass Index (BMI) was calculated by using height in centimeters and weight in kilograms.
Time Frame: Week 4 and Week 8
Measure: Mean (Standard Error); unit: BMI Kg/m2
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo - Sugar Pill
Number analyzed (Participants) | 48 | 51
BMI Kg/m2
  Baseline | 27.85 (1.0) | 27.69 (0.081)
  Week 4 | 28.14 (1.01) | 27.91 (0.84)
  Week 8 | 27.73 (0.99) | 28.04 (0.82)

ADVERSE EVENTS:
Time Frame: 56 days
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg | Placebo - Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/49 | 1/52
Other Adverse Events (participants affected / at risk) | 26/49 | 26/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg (N=49) | Placebo - Sugar Pill (N=52)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg (N=49) | Placebo - Sugar Pill (N=52)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 4 (4) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (4)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 5 (5)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other